CLINICAL TRIAL: NCT04353323
Title: Comparison of the Proportion of Covid19 Seroconversion of Caregivers Working or Not in the COVID Sector
Brief Title: COVID 19-Caregivers IGg Seroconversion
Acronym: CoSigS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20_0016/CoSigS
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Infection, COVID-19
MeSH Terms: conditions — Infections; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Covid area
  Interventions: Other: Blood sampling
- Non-Covid area
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — 3 blood samples (D0, D15 and D30) will be taken from each participant

SUMMARY:
According to recent publications, the percentage of caregivers infected with COVID 19 is evaluated between 10 and 30% . This great variability is due, on the one hand to the intensity of the influx of covid plus patients and, on the other hand, to the disparity in the preparation of caregivers in the face of this emergency. Indeed, we can understand that the strict application of hygiene rules can be faulted in the face of the volume of patients, the lack of protective equipment and the lack of specific training for caregivers in this area. As a result, within healthcare teams, there are many questions that generate anxiety: will I be able to provide care properly while protecting myself from the risk of contamination? This anxiety is also present and sometimes manifests itself aggressively in the entourage or in the vicinity of caregivers, due to lack of scientific data adapted to the local ecology of the crisis.

Thus, the aim of this study is to show that the risk for caregivers of being contaminated by COVID in an area dedicated to COVID positive patients is no higher than being a caregiver in a non-COVID area that he either in the adult or pediatric sector.

ELIGIBILITY:
Inclusion Criteria:

* caregivers staff assigned to a non-intensive care COVID service
* or caregivers staff assigned to a non-COVID adult service
* or caregivers staff assigned to a non-COVID pediatric service
* Age > = 18 years old
* With health insurance
* Express consent

Exclusion Criteria:

* Protected persons
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers staff assigned to a non-intensive care COVID service
  * Or caregiversg staff assigned to a non-COVID adult service
  * Or caregivers staff assigned to a non-COVID pediatric service
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2020-06-25 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
Seroconversion | Day1
  Participants seroconverion will be assessed by analysing IgG When the seroconverion is confirmed (whenever it occurs), the participant ends his partipation.
Seroconversion | Day 15
  Participants seroconverion will be assessed by analysing IgG When the seroconverion is confirmed (whenever it occurs), the participant ends his partipation.
Seroconversion | Day 30
  Participants seroconverion will be assessed by analysing IgG When the seroconverion is confirmed (whenever it occurs), the participant ends his partipation.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France